CLINICAL TRIAL: NCT01996657
Title: D-dimer Levels Determined the Intensity of Anticoagulation Therapy to Improve Outcomes in Patients With Mechanical Valve Replacement
Brief Title: D-Dimer Determined Anticoagulation INTENSITY in Patients With Mechanical Valve Replacement
Acronym: 3D-INTENSITY
Status: Completed | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-P-002
Record Dates: First submitted 2013-11-04; First posted 2013-11-27 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2016-06

CONDITIONS: Heart Valve Disease
Keywords: mechanical valves replacement; INR; D-dimer; thromboembolic events
MeSH Terms: conditions — Heart Valve Diseases; Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Standard intensity of anticoagulation: After mechanical valve replacement，patients should be gave oral anticoagulants，such as warfarin.and The intensity of anticoagulation for this group was standard intensity (INR:2.5-3.5).
  Interventions: Drug: Warfarin
- Low intensity and adjusted by elevated D-dimer: The intensity of anticoagulation maintained at low level initiatively, D-dimer testing were analyzed at 3 month later. In case of D-dimer level elevated, adjusted the intensity to standard level.
  Interventions: Drug: Warfarin
- Low intensity without adjustment: The intensity of anticoagulation for this group was kept at low intensity without adjustment (INR:1.8-2.6),
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin
  Other Names: Warfarin Sodium Tablets

SUMMARY:
The optimal intensity of oral anticoagulation in China patients undergoing mechanical valve replacements is still controversial due to the different risk profiles of thrombophilia and bleeding in Chinese patients. Elevated D-dimer could reflect a pro-thrombogenic or prothrombotic state, and thus might be used to decide the intensity of oral anticoagulation.

This study was to evaluate whether elevated D-dimer levels could help to determine the intensity of oral anticoagulation in patients with mechanical heart valve prostheses.

DETAILED DESCRIPTION:
Background: The optimal intensity of oral anticoagulation in China patients undergoing mechanical valve replacements is still controversial due to the different risk profiles of thrombophilia and bleeding in Chinese patients. Elevated D-dimer could reflect a pro-thrombogenic or prothrombotic state, and thus might be used to decide the intensity of oral anticoagulation.

Objective: This study was to evaluate whether elevated D-dimer levels could help to determine the intensity of oral anticoagulation in patients with mechanical heart valve prostheses.

Methods: A single-center, prospective study was performed. 748 Patients with mechanical valve replacement who had received oral anticoagulation. The patients were randomly assigned to three groups The intensity of anticoagulation for group one was standard intensity (INR:2.5-3.5). The intensity of anticoagulation for group two was kept at low intensity without adjustment (INR:1.8-2.6), and for group three , The intensity of anticoagulation maintained at low level initiatively (INR:1.8-2.6), D-dimer testing were analyzed two times at 3 month later. In case of D-dimer level elevated, adjusted the intensity of anticoagulation to standard level. The endpoint of the study was the subsequent thromboembolic and major bleeding during an average follow-up of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. age>18years,male or female without pregnancy;
2. Suffered the mechanical valves replacement in Wuhan Asia Heart Hospital;
3. The operation type was Mitral valve replacement or Double valves replacement(aortic and mitral valve replacement).

Exclusion Criteria: Patients with following diseases within 3 months.

1. deep venous thromboembolism
2. Pulmonary embolism
3. Aortic dissection
4. stroke
5. Cerebral hemorrhage
6. Myocardial infarction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffered mechanical valves replacement because of valves dysfunction; and oral anticoagulation therapy with warfarin
Sampling Method: Non-Probability Sample
Enrollment: 772 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: zhang zhenlu, PH.D, Study Director — Wuhan Asia Heart Hospital; Zhou xin, Doctor, Study Chair — Wuhan Asia Heart Hospital; liu ze jin, PH.D, Study Director — Wuhan Asia Heart Hospital
Locations (2):
- China (2):
  - WAHH, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang L, Long Y, Xiao H, Yang J, Liu X, Zhang Z. D-Dimer to Predict the Clinical Outcomes in Patients with Mechanical Heart Valve Replacement During Oral Anticoagulation Therapy. Int Heart J. 2019 May 30;60(3):631-636. doi: 10.1536/ihj.18-237. Epub 2019 Apr 25. PMID 31019170
- [Derived] Zhang L, Zheng X, Long Y, Wu M, Chen Y, Yang J, Liu Z, Zhang Z. D-dimer to guide the intensity of anticoagulation in Chinese patients after mechanical heart valve replacement: a randomized controlled trial. J Thromb Haemost. 2017 Oct;15(10):1934-1941. doi: 10.1111/jth.13782. Epub 2017 Sep 20. PMID 28762606

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Intensity of Anticoagulation: After mechanical valve replacement，patients should be gave oral anticoagulants，such as warfarin.and The intensity of anticoagulation for this group was standard intensity (INR:2.5-3.5).
  Warfarin
- Low Intensity and Adjusted by Elevated D-dimer: The intensity of anticoagulation maintained at low level initiatively, D-dimer testing were analyzed at 3 month later. In case of D-dimer level elevated, adjusted the intensity to standard level.
  Warfarin
- Low Intensity Without Adjustment: The intensity of anticoagulation for this group was kept at low intensity without adjustment (INR:1.8-2.6),
  Warfarin
Period: Overall Study
Arm/Group | Standard Intensity of Anticoagulation | Low Intensity and Adjusted by Elevated D-dimer | Low Intensity Without Adjustment
Started | 250 | 250 | 248
Completed | 237 | 239 | 234
Not Completed | 13 | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Intensity of Anticoagulation | Low Intensity and Adjusted by Elevated D-dimer | Low Intensity Without Adjustment | Total
Number analyzed (Participants) | 237 | 239 | 234 | 710
Age, Continuous [Median (Standard Deviation); unit: years] | 48.8 (11.5) | 50.4 (11.9) | 50.1 (10.9) | 49.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 102 | 96 | 311
  Male | 124 | 137 | 138 | 399
Elevated D-dimer(n) [Number; unit: participants] | 17 | 36 | 38 | 91

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Events;
Description: The bleeding events included cerebral hemorrhage, gastrointestinal bleeding and other major internal or external bleeding that causes death, hospitalization, or permanent injury (e.g. vision loss) or necessitates transfusion.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Intensity of Anticoagulation | Low Intensity and Adjusted by Elevated D-dimer | Low Intensity Without Adjustment
Number analyzed (Participants) | 237 | 239 | 234
Participants | 16 | 3 | 4

2. Primary Outcome: Thrombotic Events
Description: The thrombotic events included valve thrombosis, transient ischemic attack, ischemic stroke, peripheral embolism, and myocardial infarction.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Intensity of Anticoagulation | Low Intensity and Adjusted by Elevated D-dimer | Low Intensity Without Adjustment
Number analyzed (Participants) | 237 | 239 | 234
Participants | 5 | 5 | 14

3. Secondary Outcome: All Cause Deaths
Description: The deaths from all causes
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Intensity of Anticoagulation | Low Intensity and Adjusted by Elevated D-dimer | Low Intensity Without Adjustment
Number analyzed (Participants) | 237 | 239 | 234
Participants | 12 | 4 | 5

ADVERSE EVENTS:
Groups:
- D-dimer-guided Adjustmentd of Anticoagutlation Intensity: The intensity of anticoagulation maintained at low level initiatively, D-dimer testing were analyzed at 3 month later. In case of D-dimer level elevated, adjusted the intensity to standard level.
  Warfarin
Arm/Group | Standard Intensity of Anticoagulation | D-dimer-guided Adjustmentd of Anticoagutlation Intensity | Low Intensity Without Adjustment
All-Cause Mortality (participants affected / at risk) | 12/245 | 4/245 | 5/242
Serious Adverse Events (participants affected / at risk) | 24/245 | 9/245 | 20/242
Other Adverse Events (participants affected / at risk) | 0/245 | 0/245 | 0/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Intensity of Anticoagulation (N=245) | D-dimer-guided Adjustmentd of Anticoagutlation Intensity (N=245) | Low Intensity Without Adjustment (N=242)
thrombotic envents (Blood and lymphatic system disorders) | 5 | 5 | 14 — including valve thrombosis, transient ischemic attack, ischemic stroke, peripheral embolism, and myocardial infarction.
bleeding events (Blood and lymphatic system disorders) | 16 | 3 | 4 — including cerebral hemorrhage, gastrointestinal bleeding and other major internal or external bleeding that causes death, hospitalization, or permanent injury (e.g. vision loss) or necessitates transfusion.
Deaths from other causes (Cardiac disorders) | 3 | 1 | 2 — Death from Heart failure,Cancer or unexplained death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes